CLINICAL TRIAL: NCT05178238
Title: Intestinal Microbiota of Patients Hospitalized With Sars-CoV-2
Acronym: MICRODIGCOV
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2021-1/AS-01
Record Dates: First submitted 2021-12-18; First posted 2022-01-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
Keywords: microbiota; gastrointestinal microbiome; translocation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal and blood samples taken for a biobank
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with high viral load of SARS-CoV-2 in feces
  Interventions: Other: Fecal sample
- Patients with low viral load of SARS-CoV-2 in feces
  Interventions: Other: Fecal sample

INTERVENTIONS:
Other: Fecal sample — Fecal sample taken to investigate intestinal microbiota

SUMMARY:
The study investigators hypothesize that SARS-Cov2 infection alters the composition of the digestive microbiota and its functionality, resulting in changes in intestinal permeability and consequently in microbial digestive translocation. These changes may correlate with the magnitude of the SARS-CoV-2 viral load in the gastrointestinal tract and may have an impact on the clinical manifestations and evolvability of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized at in Nimes University hospital
* Infection with SARS-CoV-2 confirmed by RT-PCR
* The patient must have signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in an interventional study susceptible to modify the intestinal microbiota, or is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient with a chronic digestive pathology or having been operated in the previous year or having enteral nutrition or having had bariatric surgery
* Patient is pregnant, parturient or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients hospitalized in the Nimes University Hoptial with SARS-CoV-2 infection confirmed by RT-PCR
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) | Day 0
  RT-qPCR of SARS-CoV-2 to calculate copies/mg

SECONDARY OUTCOMES:
Age of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  Age in years
Sex of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  Male/female
Clinical features of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  Date of start of symptoms, current therapeutics, antibiotic therapy, blood pressure, heart rate, respiration rate, oxygen saturation, symptoms, Covid stage (ordinal 8 stage scale)
Total blood count of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
  lymphocyte count, eosinophil count
C-reactive protein level biological data of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
  concentration
Fibrinogen level of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
  concentration
Lactate Dehydrogenase of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
  concentration
D-dimer level of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
  concentration
Ferritin levels, of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
  Concentration
Albumin levels of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  concentration
Calcium levels of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
  concentration
Glomerular filtration rate of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
  volume per time
Liver function tests of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
Cytobacteriological urine exam of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
Blood cultures of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
Other infectious samples (other than SARS-CoV-2) of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) if tested | Day 0
Taxonomic features of intestinal microbiota of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  Number of Operational Taxonomic Unit
Percentage of Operational Taxonomic Units in intestinal microbiota of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  %
Diversity of intestinal microbiota of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  Shannon Index
Diversity of intestinal microbiota of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  Bray Curtis Index
LPS-binding Protein concentration of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  pg/ml ELISA
soluble CD14 concentration of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  ng/ml ELISA
RNA16s concentration of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  PCR and sequencing
RNA18 concentration of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  PCR and sequencing
I-FAB concentration of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  ng/ml:ELISA
Claudin 3 concentration of patients with high viral load of SARS-CoV-2 in feces (>50 copies/mg) versus low viral load (≤50 copies/mg) | Day 0
  ng/ml:ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Albert Sotto, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France